CLINICAL TRIAL: NCT04899297
Title: Quality of Life in Parents of Conservatively Treated Adolescents With Spinal Deformities: Development of a New Questionnaire.
Brief Title: Quality of Life in Parents of Adolescents With Spinal Deformities: Development of a New Questionnaire.
Status: Active, not recruiting | Type: Observational
Sponsor: Istituto Scientifico Italiano Colonna Vertebrale (Other)
Responsible Party: Sponsor
Other Study IDs: PQOL-Isico
Record Dates: First submitted 2021-05-06; First posted 2021-05-24 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Quality of Life; Spinal Deformity; Scoliosis; Adolescence
Keywords: Scoliosis; Quality of life; Spinal Deformity
MeSH Terms: conditions — Scoliosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Quality of life
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — All parents of patients visited at an outpatient service dedicated to the treatment of vertebral deformities will be recruited at the end of the medical clinical evaluation. The doctor will invite all subjects to complete the questionnaire anonymously at the end of each follow-up visit.

SUMMARY:
This study aims to develop a new instrument capable of providing an efficient measure of the quality of life of parents of conservatively treated patients with spinal deformity. The development of a questionnaire in a Rasch environment and specifically developed for parents of conservatively treated patients will ensure greater sensitivity and specificity of the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* have at least one child between the ages of 10 and 18 with adolescent idiopathic scoliosis of 10 degrees or more, or with Scheuermann's kyphosis or idiopathic hyperkyphosis
* prescription of a brace or specific exercises for the child's vertebral deformity.

Exclusion Criteria:

* Child with a history of spinal surgery
* Child with a history of significant diseases with possible impact on the quality of life of the parents
* Child with a history of spinal trauma
* Child with positive neurological evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parents of adolescents with spinal deformities treated in a tertiary referral outpatient center.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Parents' quality of life | through study completion, an average of 1 year
  New questionnaire developped to assess quality of life of parents of patients with spinal deformity treated conservatively

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Zaina, MD, Principal Investigator — Istituto Scientifico Italiano Colonna Vertebrale
Locations (1):
- ISICO, Milan, Mi, Italy

IPD SHARING:
Plan to Share IPD: No